CLINICAL TRIAL: NCT01234532
Title: GCC 0927 A Pilot and Phase II Study of Entinostat and Anastrozole/Tamoxifen in Women With Triple Negative Breast Cancer to Evaluate Biomarkers and Surrogates for Response
Brief Title: Entinostat and Anastrozole in Treating Postmenopausal Women With TNBC That Can Be Removed by Surgery
Acronym: 0927GCC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00047658; NCI-2011-02542 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000687507; 8597 (Other: CTEP)
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Results first posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Estrogen Receptor-negative Breast Cancer; HER2-negative Breast Cancer; Progesterone Receptor-negative Breast Cancer; Stage I Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Triple-negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — entinostat; Anastrozole; Mastectomy, Segmental; Mastectomy

STUDY DESIGN:
Intervention Model Description: no masking
Masking Description: no masking

ARMS (1):
- entinostat & anastrozole neoadjuvant (Experimental): Neoadjuvant entinostat daily on days 1, 8, 15, 22, and 29 + anastrozole daily on days 4-29 followed by surgery ie either lumpectomy or mastectomy.
  Correlative studies will be performed utilizing tissue and blood. A baseline tumor biopsy is done prior to study entry or archival tissue from diagnosis may be used and a representative tumor sample is submitted at time of surgery.
  Bloods are drawn for correlative sciences on day 1 and 15 of treatment prior to entinostat dosing and 30 mins post and again on day of surgery.
  Interventions: Drug: entinostat; Drug: anastrozole; Other: diagnostic laboratory biomarker analysis; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: entinostat — orally
  Other Names: SNDX-275; MS-275
Drug: anastrozole — Given PO
  Other Names: arimidex
Other: diagnostic laboratory biomarker analysis — Correlative studies will be performed utilizing tissue and blood. A baseline tumor biopsy is done prior to study entry or archival tissue from diagnosis may be used and a representative tumor sample is submitted at time of surgery.
  Bloods are drawn for correlative sciences on day 1 and 15 of treatment prior to entinostat dosing and 30 mins post and again on day of surgery.
Procedure: therapeutic conventional surgery — Lumpectomy or mastectomy will be performed follwoing day 29 of study therapy
  Other Names: Lumpectomy or mastectomy

SUMMARY:
This phase II trial is studying how well giving entinostat and anastrozole together works in treating postmenopausal women with triple-negative breast cancer that can be removed by surgery. Entinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Estrogen can cause the growth of breast cancer cells. Hormone therapy using anastrozole may fight breast cancer by blocking the use of estrogen by the tumor cells. Giving entinostat together with anastrozole may be an effective treatment for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of entinostat in combination with anastrozole or tamoxifen. (Pilot) II. To determine the optimal dose of entinostat in combination with anastrozole or tamoxifen for phase II. (Pilot) III. To determine baseline and percentage change in proliferative index (Ki67) before and after treatment with entinostat and anastrozole/tamoxifen in triple negative breast cancer (TNBC). (Phase II) IV. To determine the estrogen receptor (ER) expression after treatment with entinostat and anastrozole/tamoxifen in TNBC. (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate baseline and change in the expression levels of progesterone receptor (PR), human epidermal growth factor receptor 2 (HER2), epidermal growth factor receptor (EGFR), cytokeratin 5/6 (CK5/6), and aromatase before and after treatment with entinostat and anastrozole/tamoxifen.

II. To assess baseline and change in tumor tissue histone H3 and H4 acetylation before and after treatment with entinostat and anastrozole/tamoxifen.

III. To assess the clinical and pathological response to preoperative combination of entinostat and anastrozole/tamoxifen in TNBC.

TERTIARY OBJECTIVES:

I. To correlate the levels of histone H3 and H4 acetylation in tumors with the changes in Ki67 and ER.

II. To evaluate baseline and change in gene methylation silencing and expression of candidate genes in tissues and in circulating DNA, including estrogen receptor (ER)-alpha, ER-beta, RAR-beta, cyclin D2, Twist, RASSF1A, and HIN-1.

III. To correlate entinostat trough concentrations with histone H3 and H4 acetylation in tumors as well as the change in Ki67 and ER.

IV. To evaluate baseline and change in the global gene expression profile before and after treatment with entinostat and anastrozole/tamoxifen.

OUTLINE: This is a multicenter, pilot study followed by a phase II study.

Patients receive entinostat orally (PO) once daily on days 1, 8, 15, 22, and 29 and anastrozole PO once daily on days 4-29. Patients then undergo mastectomy or lumpectomy.

Tumor tissue samples are collected at baseline or from original diagnosis, and during surgery for correlative studies by IHC and RT-PCR. Blood samples are also collected at baseline, on days 1 and 15, and during surgery for correlative studies.

After completion of study therapy, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria

* Female greater than or equal to 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status <2 (see Appendix A).
* Histologically confirmed adenocarcinoma of the breast.
* Evidence of hormone insensitivity (ER and PR negative) of primary tumor tissue. ER negative is define as ER 0 or < 1% staining by immunohistochemistry. PR negativity is defined as PR < 1% staining by immunohistochemistry.
* HER2 negative in the primary tumor tissue as defined by:

  * Immunohistochemistry (IHC) Grade 0 as defined by no staining observed or membrane staining that is incomplete and is faint/barely perceptible and within ≤10% of the invasive tumor cell
  * IHC 1+ as defined by incomplete membrane staining that is faint/barely perceptible and within >10% of the invasive tumor cell
  * IHC Grade 2+ staining intensity by means of IHC analysis with no gene amplification below.
  * No gene amplification on ISH based on

    * Single-probe average HER2 copy number <4.0 signals/cell
    * Dual-probe HER2/CEP17 ratio <2.0 with an average HER2 copy number <4.0 signals/cell
* Ability to understand and the willingness to sign a written informed consent document.
* Patients must not have received any prior chemotherapy, radiation therapy, or endocrine therapy for their current breast cancer. Patients who received tamoxifen or raloxifene or another agent for prevention of breast cancer may be included as long as the patient has discontinued the treatment at least one month prior to baseline study biopsy.
* Women of childbearing potential must have negative (serum or urine) pregnancy test within 7 days prior to registration.
* Patients must have adequate tumor tissue sample prior to the enrolment available for correlative studies as defined below:

  * Core needle biopsy or incisional biopsy samples that can provide ≥ 3 unstained sections of 5 micron thickness. Fine needle aspiration (FNA) sample alone is not sufficient except in the second cohort.
  * Additional core needle biopsy needs to be performed in the patients who agree to participate in this study and do not have adequate tumor tissue sample.
* Patients must have adequate organ and marrow function as defined below:

  * Hemoglobin ≥ 9.0 g/dL
  * Leukocytes >2,500/mcL
  * Absolute neutrophil count >1,100/mcL
  * Platelets >100,000/mcL
  * Total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) <2.5 x institutional upper limit of normal
  * Creatinine within normal institutional limits or creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal

Additional Inclusion Criteria for the First cohort:

- Unresected operable breast cancer that meets the following clinical stages (see Appendix B):

* T1b, T1c, or T2
* N0 or N1
* M0 (No distant metastasis)

Additional Inclusion Criteria for the Second cohort:

* Unresectable, inoperable, recurrent local-regional breast cancer or
* Metastatic (stage IV) breast cancer
* Patients must have measurable or evaluable disease (i.e. ascites or pleural/pericardial effusion). Patients with bone metastatic only will be excluded.
* Patients must not have rapidly progressive disease, extensive visceral involvement, or any high risk characteristics that are not appropriate for this treatment as per investigator's discretion.
* Patients must receive at least one prior line of chemotherapy but not more 2 prior chemotherapy regimens for stage IV breast cancer. Prior chemotherapy in the adjuvant and /or neoadjuvant setting is permitted. However, patients must have finished chemotherapy at least 2 weeks prior to enrollment.
* Patients must have an accessible tumor lesion from which a fine needle aspirate or preferably a core biopsy specimen can be obtained. Patients with FNA only samples are allowed in this cohort. Ascites or pleural/pericardial effusion alone is not sufficient.
* Patients must be willing to provide consents for 2 research biopsies. However, the pretreatment biopsy can be omitted in patients who have recent biopsy but have not been started on breast cancer treatment within 12 weeks prior to the registration and there is adequate tumor tissue sample

Exclusion Criteria

* Patients may not be receiving any other investigational agents.
* Prior exposure to other HDAC inhibitors. However, prior valproic acid exposure is allowed providing

  ≥ 30 days wash-out period.
* History of allergic reactions or hypersensitivity to compounds of similar chemical or biologic composition to entinostat, benzamide, anastrozole, or tamoxifen.
* Any medical condition which in the opinion of the investigator puts the patient at risk of potentially serious complications while on this therapy. Examples: HIV, unstable angina, uncontrolled heart failure or hypertension, uncontrolled hyperlipidemia, uncontrolled diabetes mellitus, uncontrolled systemic infection.
* Previous or current systemic malignancy within the past 3 years other than breast cancer or adequately treated cervical carcinoma in situ or basal/squamous carcinoma of the skin.

Inclusion of Minorities

- Women of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-10; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saranya Chumsri, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Maryland Baltimore, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Entinostat & Anastrozole Neoadjuvant: Neoadjuvant entinostat daily on days 1, 8, 15, 22, and 29 + anastrozole daily on days 4-29 followed by surgery ie either lumpectomy or mastectomy.
  Correlative studies will be performed utilizing tissue and blood. A baseline tumor biopsy is done prior to study entry or archival tissue from diagnosis may be used and a representative tumor sample is submitted at time of surgery.
  Bloods are drawn for correlative sciences on day 1 and 15 of treatment prior to entinostat dosing and 30 mins post and again on day of surgery.
  entinostat: orally
  anastrozole: Given PO
  diagnostic laboratory biomarker analysis: Correlative studies will be performed utilizing tissue and blood. A baseline tumor biopsy is done prior to study entry or archival tissue from diagnosis may be used and a representative tumor sample is submitted at time of surgery.
  Bloods are drawn for correlative sciences on day 1 and 15 of treatment prior to entinostat dosing and 30 mins post and again on day of surgery.
Period: Overall Study
Arm/Group | Entinostat & Anastrozole Neoadjuvant
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Entinostat & Anastrozole Neoadjuvant: Neoadjuvant entinostat daily on days 1, 8, 15, 22, and 29 + anastrozole daily on days 4-29 followed by surgery ie either lumpectomy or mastectomy.
Arm/Group | Entinostat & Anastrozole Neoadjuvant
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 59 [48 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Dose of Entinostat in Combination With Anastrozole (Pilot)
Description: Since the study was terminated early there was insufficient data for analysis and to recommend a phase II dose of entinostat in combination with anastrozole
Time Frame: Duration of the study is 29 days followed by 30 days end of study assessment visit, up to 59 days
Population: Since the study was terminated early there was insufficient data for analysis and to recommend a phase II dose of entinostat in combination with anastrozole
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Entinostat & Anastrozole Neoadjuvant
Number analyzed (Participants) | 5
mg | NA (NA) — Data were below the lower limit of quantification

2. Primary Outcome: Number of Participants With Adverse Events
Description: To address the safety of the regimen, a maximum width 90% confidence interval for any grade 3 or higher toxicity will be approximately 30%. For 5 patients in this study, if the true unknown probability of a rare toxicity is 10%, the probability of observing 1 or more toxicities is 97%, and if the true toxicity rate is 5% then the probability of observing one or more rare toxicities is 83%.
Time Frame: Participants were followed during the study and for 30 days post treatment, up to 59 days
Measure: Count of Participants; unit: Participants
Arm/Group | Entinostat & Anastrozole Neoadjuvant
Number analyzed (Participants) | 5
Participants | 5

3. Primary Outcome: Change in Proliferative Index (Ki67) (Phase II)
Description: The 95% confidence intervals will be constructed for the observed proportions. Exploratory data analysis and appropriate graphs will be used to decide whether data transformation (e.g. log or square-root) is necessary to assure an approximate normality. All descriptive statistics will be reported for ER and Ki67 expression. The general linear model approach and/or its non parametric alternative, the Wilcoxon test, will be used to assess whether there is any evidence of changes due to treatment.
Time Frame: Baseline to the time of surgery, within 6 days after the last dose of entinostat, up to 35 days
Population: Since the study was terminated early there was insufficient data to do analysis
Measure: Number (95% Confidence Interval); unit: percentage of Ki 67 expression
Arm/Group | Entinostat & Anastrozole Neoadjuvant
Number analyzed (Participants) | 5
percentage of Ki 67 expression | NA [NA to NA] — Data were below the lower limit of quantification

4. Primary Outcome: Change in Estrogen-receptor (ER) Expression (Phase II)
Description: as for outcome 3
Time Frame: Baseline before the study treatment and at the time of surgery, up to 30 days
Population: Since the study was terminated early there was insufficient data to do the analysis
Measure: Number (95% Confidence Interval); unit: percentage of (ER) expression
Arm/Group | Entinostat & Anastrozole Neoadjuvant
Number analyzed (Participants) | 5
percentage of (ER) expression | NA [NA to NA] — Data were below the lower limit of quantification

5. Secondary Outcome: Clinical Response to Entinostat and Anastrozole
Description: Rate of clinical response % of patients responding
Time Frame: Clinical response was assessed during the study treatment and before the surgery, up to 29 days
Population: Since the study was terminated early there was insufficient data to do the analysis
Arm/Group | Entinostat & Anastrozole Neoadjuvant
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in HER2
Description: Will be treated as continuous variables. Multivariate analysis of variance may also be used to compare correlated biomarkers' expression. Correlation between biomarkers will be estimated and tested. The repeated measures model approach will be also used. Categorical outcome data (e.g., number of proteins expressed) will be recorded, proportions will be estimated and compared using the Fisher's exact test.
Time Frame: Baseline before study treatment and at the time of surgery, up to 30 days
Population: Since the study was terminated early there was insufficient data to do the analysis
Measure: Number (95% Confidence Interval); unit: score on a scale
Arm/Group | Entinostat & Anastrozole Neoadjuvant
Number analyzed (Participants) | 5
score on a scale | NA [NA to NA] — Data were below the lower limit of quantification

7. Secondary Outcome: The Pathological Response to Entinostat and Anastrozole
Description: Rate of Pathologic response % of patients responding
Time Frame: Pathological response was assessed after the surgery, up to 59 days
Population: Since the study was terminated early there was insufficient data to do the analysis and data was not collected
Arm/Group | Entinostat & Anastrozole Neoadjuvant
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year, 3 months
Description: Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Arm/Group | Entinostat & Anastrozole Neoadjuvant
All-Cause Mortality (participants affected / at risk) | 2/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entinostat & Anastrozole Neoadjuvant (N=5)
Nausea (Gastrointestinal disorders) | 2 (5) — Grade 1
Nausea (Gastrointestinal disorders) | 1 (5) — Grade 2
Acid Reflux (Gastrointestinal disorders) | 2 (5) — Grade 1
Acid Refulx (Gastrointestinal disorders) | 2 (5) — Grade 2
Fatigue (General disorders) | 2 (5) — Grade 1
Fatigue (General disorders) | 1 (5) — Grade 2
Diarrhea (Gastrointestinal disorders) | 1 (5) — Grade 1
Diarrhea (Gastrointestinal disorders) | 1 (5) — Grade 2
Hot Flashes (General disorders) | 1 (5) — Grade 1
Myalgias (Infections and infestations) | 1 (5) — Grade 3
Arhralgias (Musculoskeletal and connective tissue disorders) | 1 (5) — Grade 3

LIMITATIONS AND CAVEATS:
Study was closed due to slow accrual and was not completed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-09): https://cdn.clinicaltrials.gov/large-docs/32/NCT01234532/Prot_SAP_000.pdf